CLINICAL TRIAL: NCT00306371
Title: Comparison of Stacked-Pulses Vs. Double-Pass Treatments of Facial Acne With a 1450 Nm Laser
Status: Completed | Type: Observational
Sponsor: Skincare Physicians of Chestnut Hill (Other)
Collaborators: Candela Corporation (Industry)
Other Study IDs: 20040308; WIRB study # 1056817
Record Dates: First submitted 2006-03-22; First posted 2006-03-23 (Estimated); Last update posted 2006-03-23 (Estimated); Status verified 2004-07

CONDITIONS: Acne; Acne Scars
Keywords: diode; laser; acne; acne scar
MeSH Terms: conditions — Acne Vulgaris | interventions — Lasers, Semiconductor

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Device: 1450nm diode laser

SUMMARY:
Acne can be treated with a mid-infrared laser. We demonstrated safety and efficacy using lower energy settings in order to make the treatments less painful

DETAILED DESCRIPTION:
Numerous light based therapies are currently being used for the treatment of acne. Non-ablative mid-infrared lasers have the advantage of decreasing inflammatory acne and improving acne scars. Specifically, the 1450 nm laser has been shown to be quite effective. However, it is associated with considerable pain at higher fluences despite topical anesthetics, especially when treating inflammatory acne. The goal of this study was to determine the possibility of using low fluence settings to treat moderate to severe acne at a more tolerable pain level without compromising treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* acne lesion count of at least 10 inflammatory papules on each side of the face and a severity grade consistent with color photographs in the Allen & Smith grading scale of greater than or equal to grade 3 and no worse than grade 5

Exclusion Criteria:

* Exclusion criteria included the use of oral retinoids or systemic corticosteroids within the past 6 months and the use of all prescription topical or systemic anti-acne medications 4 weeks prior to the initiation of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2004-07; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: Nathan S Uebelhoer, DO, Principal Investigator — Skincare Physicians of Chestnut Hill; Jeffrey S Dover, MD, Study Director — Skincare Physicians of Chestnut Hill; Kenneth A Arndt, MD, Study Chair — Skincare Physicians of Chestnut Hill
Locations (1):
- Skincare physicians of Chestnut Hill, Chestnut Hill, Massachusetts, United States